CLINICAL TRIAL: NCT06624462
Title: Effectiveness of a Pragmatic, Metabolic Care Clinic for Patients With Severe Mental Illness - The Meta Care Clinic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bjorn H. Ebdrup (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); University of Toronto (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Sponsor-Investigator, Bjorn H. Ebdrup, MD, consultant, PhD and clinical professor in psychiatry Bjørn Hylsebeck Ebdrup, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The Meta Care Clinic; H-23045618 (Other: Scientific Ethics Committees for the Capital Region of Denmark); p-2023-14342 (Other: The Danish Data Protection Agency); 2096-00099B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2024-09-04; First posted 2024-10-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Severe Mental Disorder; Metabolic Complication; Side-Effect;Medication; Schizophrenia Spectrum and Other Psychotic Disorders; Bipolar Disorder
Keywords: Severe mental illness; Overweight and obesity; Antipsychotic medication; Dysmetabolism; Schizophrenia Spectrum Disorders; Bipolar disorder
MeSH Terms: conditions — Mental Disorders; Drug-Related Side Effects and Adverse Reactions; Schizophrenia Spectrum and Other Psychotic Disorders; Bipolar Disorder; Overweight; Obesity | interventions — Therapeutics; Standard of Care

STUDY DESIGN:
Intervention Model Description: Pragmatic, open label, non-blinded randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment in the Meta Care Clinic (Active Comparator): The patients who after randomization are allocated to the treatment arm will receive 12 months of treatment in a pragmatic metabolic clinic. Patients will receive measurements/monitoring at least 3 times during the study period: Upon enrolment, after 6 months and after 12 months.
  Interventions: Other: Treatment in the Meta Care Clinic
- Standard care with general practitioner and/or outpatient clinics (Active Comparator): The patients who after randomization are allocated for standard care will continue with their current psychiatric out-patient clinic and/or contact with their general practitioner. Patients will receive measurements/monitoring upon enrolment and after 12 months.
  Interventions: Other: Standard care with general practitioner and/or outpatient clinics

INTERVENTIONS:
Other: Treatment in the Meta Care Clinic — * Consultations by medical doctors with specific metabolic training from the metabolic clinic located at Centre for Addiction and Mental Health in Toronto, Canada, and an exercise physiologist.
  * Evaluation of their psychopharmacotherapy with consultation and detailed recommendations to the patients' treating psychiatrist and/or general practitioner regarding dosage reductions or switching of psychotropics if this is clinically feasible to reduce the metabolic burden.
  * Lifestyle interventions
  * Pharmacotherapy with evidence to support use to mitigate antipsychotic-induced weight gain
  * Treatment of other cardiovascular risk factors such as dyslipidaemia, hypertension, smoking and diabetes in close collaboration with recognized specialists in endocrinology.
  * Assessment of plans at conferences with participation of the sponsor, the primary investigator as well as recognized specialists in endocrinology and psychiatry.
  * Qualitative interviews will be conducted post-intervention.
  Arms: Treatment in the Meta Care Clinic
Other: Standard care with general practitioner and/or outpatient clinics — Following measurements after 12 months, patients will receive individualized lifestyle recommendations from an exercise physiologist and a MD will offer to send recommendations regarding the following potential post-trial interventions to the patients' general practitioner and/or outpatient clinic prepared in close collaboration with recognized specialists in psychiatry and endocrinology:
  * Suggestions regarding relevant psychotropic medication adjustments or switches if this is found relevant and clinically feasible to reduce the metabolic burden.
  * Suggestions regarding potential add-on of weight reducing pharmacotherapy.
  * Suggestions regarding pharmacological treatment of other cardiovascular risk factors such as dyslipidaemia, hypertension, smoking and type 2 diabetes.
  Arms: Standard care with general practitioner and/or outpatient clinics

SUMMARY:
This study will examine the effectiveness of a Pragmatic, Metabolic Care Clinic for Patients With Severe Mental Illness

DETAILED DESCRIPTION:
Severe mental illness (SMI), including schizophrenia spectrum disorders and bipolar disorder, is associated with high mortality rates and cardiovascular disease. Obesity and dysmetabolism caused by antipsychotic medication comprise modifiable risk factors, which remain undertreated.

The investigators will address the gaps in cardiometabolic care of SMI patients by examining the effectiveness of a pragmatic metabolic care clinic for patients with SMI. Moreover, the investigators will include qualitative investigation of patients' perspectives in relation to acceptability, satisfaction with care, and motivation for health behaviour change.

A total of 84 patients between 18-45 years with diagnoses of schizophrenia spectrum disorders or bipolar disorder will be recruited from inpatient and outpatient clinics in the Mental Health Services of the Capital Region of Denmark. Eligible patients are antipsychotics-treated and present with a 5% weight increase / 5 cm waistline increase since initiation of antipsychotic therapy or body mass index (BMI) ≥30 kg/m2 or BMI ≥27 kg/m2 and concomitant prediabetes, diabetes, hypertension, sleep apnoea and/or dyslipidaemia.

Patients will be enrolled in an open-label randomized controlled parallel-group trial with an allocation-ratio of 1:1 to a pragmatic, specialized metabolic clinic with measurement-based care and evidence-based best-practice treatment or standard care. The primary outcome is the proportion of patients in the intervention group achieving a weight loss ≥5% of initial body weight vs the standard care group at 12 months. Secondary and exploratory outcomes include changes in other cardiovascular risk factors, quality of life, personal recovery and cognitive measures. Finally, qualitative interviews will explore patient experience and contextual factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia spectrum disorders (International classification of diseases; ICD-10: DF2x) or bipolar disorder (ICD-10: DF30.x or DF31.x)
* Medical treatment with antipsychotics
* Age 18-45 years
* Legally competent
* Able to give informed consent

and either:

- Body mass index (BMI) ≥30 kg/m2.

Or

* BMI ≥27 kg/m2 and at least one of the following:
* Hypertension defined as treatment with ≥1 antihypertensive drug or out-of-office / 24-hour, non-invasive ambulatory blood pressure ≥140/90 mmHg within the previous 6 months
* Dyslipidaemia defined as treatment with ≥1 lipid-lowering drug or elevated low-density lipoprotein (LDL) cholesterol (≥3.0 mmol/l), elevated triglycerides (≥1.7 mmol/l) or low high-density lipoprotein cholesterol (≥1.2 mmol/l in women and ≥1.0 mmol/l in men) within the previous 6 months
* Sleep apnoea (ICD-10 DG473).
* Prediabetes or diabetes defined as HbA1c ≥42 mmol/mol or impaired fasting glucose as defined by the International Diabetes Federation within the previous 6 months.

Or

- a history of rapid weight gain during antipsychotic therapy defined as increases of either ≥5% body weight or ≥5 cm waist circumference since initiation of antipsychotic therapy.

Exclusion Criteria:

* Clinical or laboratory evidence of comorbid medical disease not compatible with participation as judged by the research team.
* Unstable psychiatric disorder as judged by the research team.
* Severe current drug or alcohol misuse as judged by the research team.
* Acute suicidal risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a weight loss of ≥5% of initial body weight. | 12 months
  Proportion of patients in the intervention group achieving a weight loss of ≥5% of initial body weight vs the standard care group at 12 months.

SECONDARY OUTCOMES:
The metabolic composite score | 12 months
  The metabolic composite score consisting of minimally 0 points and maximally five points (one point per composite; elevated waist circumference, elevated triglycerides, blood pressure, fasting plasma glucose, and reduced high-density lipoprotein), according to the definition and cut-off values of metabolic syndrome by the International Diabetes Federation. A higher score means worse outcomes. Effect measurements: differences in percentage achieving reduction of ≥1 points between groups at 12 months.
Cardiovascular risk factors | 12 months
  Cardiovascular risk factors as defined below.
Proportion of patients achieving a weight loss of ≥10% of initial body weight. | 12 months
  Proportion of patients in the intervention group achieving a weight loss of ≥10% of initial body weight vs the standard care group at 12 months.
Proportion of patients achieving a ≥50% reduction of low-density lipoprotein cholesterol | 12 months
  Proportion of patients in the intervention group achieving a ≥50% reduction of initial low-density lipoprotein cholesterol vs the standard care group at 12 months.
Body weight | 12 months
  Absolute and relative changes in body weight. Effect measurements: differences in mean changes between groups at 12 months.
Waist circumference | 12 months
  Absolute and relative changes in waist circumference. Effect measurements: differences in mean changes between groups at 12 months.
Body mass index | 12 months
  Changes in body mass index (BMI) where weight and height will be combined to report BMI in kg/m^2. Effect measurements: differences in mean changes between groups at 12 months.
Glucose | 12 months
  Fasting plasma glucose. Effect measurements: differences in mean changes between groups at 12 months.
Insulin | 12 months
  Fasting Plasma insulin. Effect measurements: differences in mean changes between groups at 12 months.
The homeostatic Model Assessment for Insulin Resistance | 12 months
  The homeostatic Model Assessment for Insulin Resistance (HOMA-IR) measured using fasting plasma glucose and fasting plasma insulin.
  Effect measurements: differences in mean changes between groups at 12 months.
Total cholesterol | 12 months
  Fasting plasma total cholesterol. Effect measurements: differences in mean changes between groups at 12 months.
Low-density lipoprotein cholesterol | 12 months
  Fasting plasma Low-density lipoprotein (LDL) cholesterol. Effect measurements: differences in mean changes between groups at 12 months.
High-density lipoprotein cholesterol | 12 months
  Fasting plasma high-density lipoprotein (HDL) cholesterol. Effect measurements: differences in mean changes between groups at 12 months.
Very Low-density lipoprotein cholesterol | 12 months
  Fasting plasma Very Low-density lipoprotein (VLDL) cholesterol. Effect measurements: differences in mean changes between groups at 12 months.
Triglycerides | 12 months
  Fasting plasma triglycerides. Effect measurements: differences in mean changes between groups at 12 months.
Heart rate | 12 months
  Resting heart rate. Effect measurements: differences in mean changes between groups at 12 months.
Blood pressure | 12 months
  Clinic blood pressure. Effect measurements: differences in mean changes between groups at 12 months.
Hemoglobin A1c | 12 months
  Hemoglobin A1c (HbA1c). Effect measurements: differences in mean changes between groups at 12 months.

OTHER OUTCOMES:
Cardiorespiratory fitness | 12 months
  Cardiorespiratory fitness assessed by the submaximal Ekblom-Bak test on a mechanically braked cycle ergometer. Effect measurements: differences in mean changes between groups at 12 months.
Body composition: Total body fat percentage | 12 months
  Total body fat percentage measured with a bioelectrical impedance analysis. Effect measurements: differences in mean changes between groups at 12 months.
Body composition: Visceral adipose tissue | 12 months
  Visceral adipose tissue measured with a bioelectrical impedance analysis. Effect measurements: differences in mean changes between groups at 12 months.
Body composition: Skeletal muscle mass. | 12 months
  Skeletal muscle mass measured with a bioelectrical impedance analysis. Effect measurements: differences in mean changes between groups at 12 months.
Personal recovery - The Brief INSPIRE Measure of Staff Support for Personal Recovery. | 12 months
  The Brief INSPIRE Measure of Staff Support for Personal Recovery. Effect measurements: differences in mean changes between groups at 12 months.
Personal recovery - The Questionnaire about the Process of Recovery. | 12 months
  The Questionnaire about the Process of Recovery (QPR). Effect measurements: differences in mean changes between groups at 12 months.
Quality of life - the World Health Organization-5 Well-being index. | 12 months
  The World Health Organization (WHO)-5 Well-being index. Effect measurements: differences in mean changes between groups at 12 months.
Cognition - The Symbol Digit Modalities Test (SDMT). | 12 months
  The Symbol Digit Modalities Test (SDMT). Effect measurements: differences in mean changes between groups at 12 months.
Cognition - The Brief Cognitive Assessment Tool in Schizophrenia | 12 months
  The Brief Cognitive Assessment Tool in Schizophrenia (B-CATS) comprised of the following:
  1. The Trail Making Test.
  2. The Letter-Number Span Record Form.
  3. The Category Fluency Test.
  Effect measurements: differences in mean changes between groups at 12 months.
Smoking Cessation | 12 months
  Smoking cessation amongst persons who are smoking at baseline measured as self-reported cessation for the past 7 days after 12 months. Effect measurements: differences in mean changes between groups at 12 months.
Physical activity | 12 months
  Physical activity of weekly self-perceived volumes of different intensities and average daily sedentary hours measured with the International Physical Activity Questionnaire. Effect measurements: differences in mean changes between groups at 12 months
Appetite | 12 months
  Appetite measured with a digital visual analogue scale (VAS) before the first meal at date of baseline measurements and date of measurements after 12 months as minimum 1 and maximally 10 with higher outcomes depicting more appetite. Effect measurements: differences in mean changes between groups at 12 months.
Qualitative evaluation | Time from study start to dropout or 12 months
  Semi-structured interviews will be conducted following the intervention with patients, who dropped out or completed the intervention, respectively. Patients who complete the intervention will be sampled purposefully to ensure maximum variation in terms of gender, age, and diagnosis, whereas the investigators will interview every patient dropping out (i.e., convenience sampling). Interviews will focus on satisfaction with the delivered care, and sustained motivation for health behaviour change. Data will be analysed by means of inductive-deductive thematic analysis informed by the COM-B model identifying capability, opportunity, and motivation as key factors which need to change in order for a behaviour change intervention to be effective. Adequate sample size for the qualitative evaluation will be guided by information power (also denoted saturation).

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn H. Ebdrup, MD, Consultant,PhD, Professor,, Study Chair — Centre for Neuropsychiatric Schizophrenia Research, CNSR, Mental Health Centre Glostrup | University of Copenhagen
Locations (1):
- Centre for Neuropsychiatric Schizophrenia Research, CNSR, Mental Health Centre Glostrup, Glostrup Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Aggregated deidentified data is expected to be available after publication upon request.